CLINICAL TRIAL: NCT03676504
Title: Treatment of Patients With Relapsed or Refractory CD19+ Lymphoid Disease With T Lymphocytes Transduced by RV-SFG.CD19.CD28.4-1BBzeta Retroviral Vector - a Unicenter Phase I/II Clinical Trial
Brief Title: Treatment of Patients With Relapsed or Refractory CD19+ Lymphoid Disease With T Cells Expressing a Third-generation CAR
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Prof. Dr. Michael Schmitt, Head of the GMP Core Facility University Hospital Heidelberg, Principal Investigator, Clinical Professor for Cellular Immunotherapy, University Hospital Heidelberg
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HD-CAR-1
Record Dates: First submitted 2018-09-07; First posted 2018-09-18 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Acute Lymphoblastic Leukemia, Adult; Acute Lymphoblastic Leukemia, Pediatric; Chronic Lymphocytic Leukemia; Diffuse Large B Cell Lymphoma; Follicular Lymphoma; Mantle Cell Lymphoma
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, Mantle-Cell | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Stratum I (Experimental): Adult patients with relapsed or refractory ALL
  Interventions: Biological: CD19.CAR T Cells; Drug: Fludarabine; Drug: Cyclophosphamide
- Stratum II (Experimental): Adult patients with relapsed or refractory CLL, DLBCL, FL or MCL
  Interventions: Biological: CD19.CAR T Cells; Drug: Fludarabine; Drug: Cyclophosphamide
- Stratum III (Experimental): Pediatric patients with relapsed or refractory ALL
  Interventions: Biological: CD19.CAR T Cells; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: CD19.CAR T Cells — Dose Level 1: 1×10^6 transduced cells/m^2; Dose Level 2: 5×10^6 transduced cells/m^2; Dose Level 3: 20×10^6 transduced cells/m^2; Dose Level 4: 5x10^7 transduced cells/m^2; Dose Level 5: 10x10^7 transduced cells/m^2; Dose Level 6: 20x10^7 transduced cells/m^2
Drug: Fludarabine — 3 days of fludarabine 30 mg/m^2/day
Drug: Cyclophosphamide — 3 days of cyclophosphamide 500 mg/m^2/day

SUMMARY:
Adult patients with r/r acute lymphoblastic leukemia (ALL) (stratum I), r/r Non-Hodgkin's lymphoma (NHL) including chronic lymphocytic leukaemia (CLL), diffuse large B-cell lymphoma (DLBCL), follicular lymphoma (FL) or mantle cell lymphoma (MCL) (stratum II) as well as paediatric patients with r/r ALL (stratum III) will be treated with autologous T-lymphocytes transduced by the third-generation RV-SFG.CD19.CD28.4-1BBzeta retroviral vector. The main purpose of this study is to evaluate safety and feasibility of escalating CD19.CAR T cell doses (0,1-20×20^7 transduced cells/m^2) after lymphodepletion with fludarabine and cyclophosphamide.

ELIGIBILITY:
Inclusion Criteria:

Stratum I/II (Adults):

* Confirmed CD19+ ALL, CLL, DLBCL, FL or MCL in patients ≥ 18 years
* ALL (Ph+ and Ph-): Confirmed CD19+ ALL by cytology and flow cytometry (FACS) AND
* Relapsed or refractory disease (including "molecular relapse" with minimal residual disease (MRD) levels > 10^-3 at two occasions > 2 weeks apart) with confirmed CD19 expression on malignant cells in relapse

  * Any relapse after allogeneic stem cell transplantation (alloSCT) (≥ 6 months from alloSCT at time of CAR T cell infusion) OR
  * Any relapse failing to achieve an MRD level of < 10^-3 after ≥ 2 lines of treatment OR
  * Primary refractory as defined by not achieving a complete remission (CR) after ≥ 2 lines of treatment
* CLL/NHL: Confirmed CD19+ CLL/NHL (including CLL, DLBCL, FL or MCL) with

  * CLL in need of treatment with:

    1. Early relapse (within 2 years) after end of chemoimmunotherapy or chemoimmunotherapy refractoriness plus failure or intolerance of both Bruton's tyrosine kinase Inhibitor (BTKi) and B-cell lymphoma 2 inhibitors (BCL-2i) OR
    2. Relapse after alloSCT, ineligible for or refractory to standard interventions (donor lymphocyte infusions (DLI), CD20 antibodies, chemoimmunotherapy)
  * DLBCL with:

    1. Refractoriness to a 2nd or later line of chemoimmunotherapy OR
    2. Relapse after autologous stem cell transplantation (autoSCT) plus ineligibility for alloSCT (including refractoriness to one line of salvage chemoimmunotherapy) OR
    3. Relapse after alloSCT
  * FL in need of treatment with:

    1. Relapse <2 years after chemoimmunotherapy AND ineligibility for or failure of autologous stem cell transplantation (autoSCT) AND ineligibility for or failure of idelalisib OR
    2. Relapse after alloSCT, ineligible for or refractory to standard interventions (DLI, CD20 antibodies, chemoimmunotherapy)
  * MCL with:

    1. Relapse after standard first-line therapy AND ineligibility for or failure to BTKi salvage therapy OR
    2. Relapse after alloSCT AND ineligibility for or failure to BTKi salvage therapy
* Measurable disease/MRD at time of enrollment
* Life expectancy ≥ 12 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 at the time of screening
* Adequate organ function:

  * Renal function defined as: serum creatinine of ≤ 2 x ULN or estimated glomerular filtration rate (eGFR) ≥ 30 mL/min/1.73 m^2
  * Liver function defined as:
  * ALT ≤ 5 times the ULN for the respective age
  * Bilirubin ≤ 2.0 mg/dl with the exception of patients with hyperbilirubinemia explained by Gilbert-Meulengracht syndrome (may be included if total bilirubin is ≤ 3.0 x ULN and direct bilirubin ≤ 1.5 x ULN) or extrahepatic disease (e.g. chronic hemolytic anemia)
  * minimum level of pulmonary reserve defined as ≤ grade 1 dyspnea and pulse oxygenation > 90% on room air
  * Hemodynamic stability and left ventricular ejection fraction (LVEF) ≥ 40% as confirmed by echocardiogram
  * Absolute neutrophil count (ANC) ≥ 500/mm3
  * Absolute lymphocyte count (ALC) ≥ 100/mm3
* Women of child-bearing potential (defined as all women physiologically capable of becoming pregnant) and all male participants must agree to use highly effective methods of contraception for one year following CD19.CAR T cell therapy
* Ability to understand the nature of the trial and the trial related procedures
* Written informed consent must be obtained prior to any screening procedures

Stratum III (Children and Adolescents with ALL):

* Age of > 3 years until < 18 years at the time of screening
* CD19+ ALL (Ph+ and Ph-) confirmed by cytology and flow cytometry (FACS) AND
* Relapsed or refractory disease (including "molecular relapse" with polymerase chain reaction (PCR) MRD > 10^-3 at two occasions > 2 weeks apart) with confirmed CD19 expression on malignant cells in relapse

  * Any relapse after alloSCT (≥ 6 months from alloSCT at time of CAR T cell infusion) OR
  * Any relapse failing to achieve an MRD level of < 10^-3 after ≥ 2 lines of treatment OR
  * Primary refractory as defined by not achieving a CR after ≥ 2 lines of treatment
* Measurable disease/MRD at time of enrollment
* Life expectancy ≥ 12 weeks
* ECOG performance status ≤ 2 (age ≥ 16 years) or Lansky performance status ≥ 50 (age < 16 years) at the time of screening
* Adequate organ function:

  * Renal function defined as serum creatinine-clearance ≥ 30 mL/min/1.73 m^2
  * Liver function defined as:
  * ALT ≤ 5 times the ULN for the respective age
  * Bilirubin ≤ 2.0 mg/dl with the exception of patients with hyperbilirubinemia explained by Gilbert-Meulengracht syndrome or extrahepatic disease (e.g. chronic hemolytic anemia)
  * minimum level of pulmonary reserve defined as ≤ grade 1 dyspnea and pulse oxygenation > 90% on room air
  * Hemodynamic stability and LVEF ≥ 40% or shortening fraction > 29% as confirmed by echocardiogram
  * ANC) ≥ 500/mm3
  * ALC ≥ 100/mm3
* Women of child-bearing potential (defined as all women physiologically capable of becoming pregnant) and postpubertal male participants must agree to use highly effective methods of contraception for one year following CD19.CAR T cell therapy
* Written informed consent of the study patient and/or the legal representative must be obtained prior to any screening procedures

Exclusion Criteria:

Stratum I/II (Adults):

* The following medications are excluded:

  * Immunosuppressive medication with the exception of ≤ 30 mg prednisolone/d or equivalent at the time of CAR T cell transfusion
  * Bridging/maintenance therapy including chemo- and immunotherapy must be stopped ≥ 2 weeks prior to leukapheresis, but can be continued between leukapheresis and lymphodepletion
* Intrathecal chemotherapy is possible at any time, but not during lymphodepletion until 14 days after CD19.CAR T cell transfusion
* Any DLI must be completed > 6 weeks prior to CD19.CAR T cell infusion
* Florid/acute or chronic Graft-versus-Host disease (GvHD)
* Uncontrolled active hepatitis B or C
* HIV-positivity
* Uncontrolled acute life-threatening bacterial, viral or fungal infection
* Severe concomitant disease (e.g. uncontrolled arterial hypertension, heart failure New York Heart Association (NYHA) III-IV, uncontrolled diabetes mellitus, uncontrolled hyperlipidemia)
* Unstable angina and/or myocardial infarction within 3 months prior to screening
* Any previous or concurrent malignancy.

The following exceptions do NOT constitute exclusion criteria:

* Adequately treated basal cell or squamous cell carcinoma (adequate wound healing is required prior to study entry)
* In situ carcinoma of the cervix or breast, treated curatively without evidence of recurrence ≥ 3 years prior to the study
* CLL or FL transformed into an aggressive B cell lymphoma
* A primary malignancy which is in complete remission for ≥ 5 years

  * Pregnant or nursing (lactating) women
  * Intolerance to the excipients of the cell product
  * Active central nervous System (CNS) involvement in ALL patient at the time of screening is not an exclusion criterion, but patients with CNS 3 status at clinical screening (d-14) are not eligible for CD19.CAR T cell transfusion
  * Participation in another clinical trial at the time of screening

Stratum III (Children and Adolescents with ALL):

* The following medications are excluded:

  * immunosuppressive medication with the exception of < 0.5 mg/d*kg body weight (BW) prednisolone-equivalent at the time of CD19.CAR T cell transfusion
  * Bridging/Maintenance therapy including chemo- and immunotherapy must be stopped ≥ 2 weeks prior to leukapheresis, but can be continued between leukapheresis and lymphodepletion
* Intrathecal chemotherapy is possible at any time, but not during lymphodepletion until 14 days after CD19.CAR T cell transfusion
* Any DLI must be completed > 6 weeks prior to CD19.CAR T cell infusion
* Florid/acute or chronic GvHD
* Uncontrolled active hepatitis B or C
* HIV-positivity
* Uncontrolled acute life-threatening bacterial, viral or fungal infection
* Severe concomitant disease (e.g. any life-limiting genetic disorder). Patients with Down Syndrome will not be excluded.
* Any previous or concurrent malignancy.

The following exceptions do not constitute exclusion criteria:

* Lymphoblastic lymphoma transformed into a CD19+ acute lymphoblastic leukemia
* A primary malignancy which is in complete remission for ≥ 5 years

  * Pregnant or nursing (lactating) women
  * Intolerance to the excipients of the cell product
  * Active CNS involvement at the time of screening is not an exclusion criterion, but patients with CNS 3 status at clinical screening (d-14) are not eligible for CD19.CAR T cell transfusion
  * Participation in another clinical trial at the time of screening

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2018-09-07 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety of CD19.CAR T cell administration assessing grade and frequency of toxicities including cytokine release syndrome (CRS) and neurotoxicity according to Common Toxicity Criteria for Adverse Events (CTCAE) | Up to 90 days after CD19.CAR T cell administration
Feasibility of CD19.CAR T cell manufacturing assessing the number of transduced T cells | Within 45 days prior to CD19.CAR T cell administration

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. Michael Schmitt, Principal Investigator — University Hospital Heidelberg, Department V; Prof. Dr. Andreas Kulozik, Principal Investigator — University Hospital Heidelberg, University Medical Center for Children and Adolescents
Locations (1):
- University Hospital Heidelberg, Heidelberg, Germany

REFERENCES:
- [Derived] Derigs P, Schubert ML, Dreger P, Schmitt A, Yousefian S, Haas S, Rothemeier C, Neuber B, Huckelhoven-Krauss A, Bruggemann M, Bernhard H, Kobbe G, Lindemann A, Rummel M, Michels B, Korell F, Ho AD, Muller-Tidow C, Schmitt M. Third-generation anti-CD19 CAR T cells for relapsed/refractory chronic lymphocytic leukemia: a phase 1/2 study. Leukemia. 2024 Nov;38(11):2419-2428. doi: 10.1038/s41375-024-02392-7. Epub 2024 Aug 27. PMID 39192036
- [Derived] Schubert ML, Schmitt A, Huckelhoven-Krauss A, Neuber B, Kunz A, Waldhoff P, Vonficht D, Yousefian S, Jopp-Saile L, Wang L, Korell F, Keib A, Michels B, Haas D, Sauer T, Derigs P, Kulozik A, Kunz J, Pavel P, Laier S, Wuchter P, Schmier J, Bug G, Lang F, Gokbuget N, Casper J, Gorner M, Finke J, Neubauer A, Ringhoffer M, Wolleschak D, Bruggemann M, Haas S, Ho AD, Muller-Tidow C, Dreger P, Schmitt M. Treatment of adult ALL patients with third-generation CD19-directed CAR T cells: results of a pivotal trial. J Hematol Oncol. 2023 Jul 22;16(1):79. doi: 10.1186/s13045-023-01470-0. PMID 37481608
- [Derived] Schubert ML, Schmitt A, Sellner L, Neuber B, Kunz J, Wuchter P, Kunz A, Gern U, Michels B, Hofmann S, Huckelhoven-Krauss A, Kulozik A, Ho AD, Muller-Tidow C, Dreger P, Schmitt M. Treatment of patients with relapsed or refractory CD19+ lymphoid disease with T lymphocytes transduced by RV-SFG.CD19.CD28.4-1BBzeta retroviral vector: a unicentre phase I/II clinical trial protocol. BMJ Open. 2019 May 19;9(5):e026644. doi: 10.1136/bmjopen-2018-026644. PMID 31110096